CLINICAL TRIAL: NCT06307548
Title: Image Guided Surgery Followed by Intraoperative Photodynamic Therapy for Improving Local Tumor Control in Patients With Loco-Regionally Advanced or Recurrent Colorectal Cancer Undergoing Surgery - Phase I/II
Brief Title: Fluorescence Image Guided Surgery Followed by Intraoperative Photodynamic Therapy for Improving Local Tumor Control in Patients With Locally Advanced or Recurrent Colorectal Cancer
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: drug shortage
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-3670923; NCI-2024-01256 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-3670923 (Other: Roswell Park Cancer Institute); UL1TR001412 (NIH)
Record Dates: First submitted 2024-02-27; First posted 2024-03-13 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Locally Advanced Colorectal Carcinoma; Recurrent Colorectal Carcinoma; Stage III Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Aminolevulinic Acid; Specimen Handling; Magnetic Resonance Spectroscopy; Photochemotherapy; 1-phenyl-3,3-dimethyltriazene; Phototherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (aminolevulinic, fluorescence-guided surgery, PDT) (Experimental): Patients receive aminolevulinic acid PO 2 to 4 hours prior to SOC surgery. Patients then undergo image-guided fluorescence 5-10 minutes post surgery, and intraoperative PDT 15-45 minutes post surgery. Patients also undergo CT or MRI during screening and on follow up. Patients also undergo blood sample collection throughout the trial.
  Interventions: Drug: Aminolevulinic Acid; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Fluorescence-Guided Surgery; Procedure: Magnetic Resonance Imaging; Drug: Photodynamic Therapy; Procedure: Surgical Procedure

INTERVENTIONS:
Drug: Aminolevulinic Acid — Given PO
  Other Names: 5-ALA; 5-Aminolaevulinic Acid; 5-Aminolevulinic Acid; Amino-Levulinic Acid; Delta Aminolevulinic Acid; Delta-Aminolevulinic Acid
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Procedure: Fluorescence-Guided Surgery — Undergo fluorescence-guided surgery
  Other Names: Fluorescence-Guided Surgical Procedure
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Photodynamic Therapy — Undergo PDT
  Other Names: PDT; Photoradiation Therapy
Procedure: Surgical Procedure — Undergo surgery
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery

SUMMARY:
This phase I/II trial studies the side effects and how well fluorescence image guided surgery followed by intraoperative photodynamic therapy for improving local tumor control in patients with colorectal cancer that has spread to nearby tissue or lymph nodes (locally advanced) or that has come back after a period of improvement (recurrent). Fluorescence image guided surgery uses a drug named aminolevulinic acid hydrochloride. Aminolevulinic acid hydrochloride is a photosensitizing agent, meaning that is activated by light and, is converted to another drug in cancer cells more than in normal cells. The converted drug emits fluorescence red light when activated with low power blue light. It is used to assist the surgeon to see cancer cells and small cancerous tissue that may have been missed during routine surgery. In addition to emitting fluorescence light, the converted drug in the cancer cells and tissue can be activated with red laser light to kill cancer cells. This procedure is called photodynamic therapy (PDT). Performing fluorescence image guided surgery followed by intraoperative photodynamic therapy after the surgical removal of the colorectal tumor before the surgical site will be closed may be effective and improve outcomes in patients with locally advanced or recurrent colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* To test the accuracy of image-guided fluorescence to detect residual disease. (Phase I)
* To determine the safety of intraoperative PDT after fluorescence-guided surgery in patients with loco-regionally advanced or recurrent colorectal cancer undergoing surgery. (Phase I)
* To determine the potential efficacy of intraoperative PDT (after image-guided fluorescence surgery). (Phase II)

SECONDARY OBJECTIVES:

* To assess the relationship between disease free survival and changes in levels of carcinoembryonic antigen (CEA) and circulating tumor DNA (ctDNA). (Phase II)
* To assess rate of recurrence by using standard-of-care computed tomography (CT) and/or magnetic resonance imaging (MRI). (Phase II)

OUTLINE:

Patients receive aminolevulinic acid orally (PO) 2 to 4 hours prior to standard of care (SOC) surgery. Patients then undergo image-guided fluorescence 5-10 minutes post surgery, and intraoperative PDT 15-45 minutes post surgery. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) during screening and on follow up. Patients also undergo blood sample collection throughout the trial.

After completion of study treatment, patients are followed up at 3 months, 24 weeks, and every 3 to 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Patients with locally advanced or recurrent colorectal cancer undergoing surgery
* Amenable to diagnostic CT and MR imaging
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 3
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Pregnant or nursing female participants
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to receive the fluorescence-guided surgery with intraoperative PDT
* Patients with porphyria, or with known hypersensitivity to porphyrins or porphyrin-like compounds
* Patients who are not cleared to undergo surgery
* Patients with any acute hepatitis or chronic liver dysfunction with baseline elevated liver function tests (i.e. Aspartate transaminase (AST)/alanine transaminase (ALT) ≥ 2.5 x upper limit of normal [ULN]) will be excluded from the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug and/or procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the fluorescence imaging (Phase I) | Up to 3 years
  Will be determined by histopathology by examining the number of true positive fluorescence cases out of the total positive fluorescence biopsies collected in the study. This will be determined by reviewing the pathology reports. The proportion of surgical cases exhibiting a positive fluorescence signal by utilizing a simple proportion along with a 95% confidence interval.
Incidence of adverse events (Phase I) | Up to 30 days post-therapy
  Will be measured by recording Gleolan administration and intraoperative photodynamic therapy (PDT) treatment related adverse events that are ≥ grade 3 with attribution of 'probable', or 'definite', according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0, that do not resolve within 7 days.
Evidence of disease (Phase II) | At 12 weeks post treatment
  Will be assessed by standard-of-care computed tomography (CT) and/or magnetic resonance imaging (MRI). The recurrence proportion and exact 95% confidence interval will be calculated.
Changes in carcinoembryonic antigen (CEA) and circulating tumor deoxyribonucleic acid (ctDNA) (Phase II) | Within 4 weeks prior to surgical/PDT intervention and 4-6 weeks after treatment
  Will be evaluated by collecting peripheral blood samples. The mean and a 95% confidence interval will be calculated around the mean change from baseline.

SECONDARY OUTCOMES:
Changes in CEA and ctDNA (Phase I) | At 4 weeks prior to surgical/PDT intervention and 4-6 weeks after treatment
  Will be evaluated by collecting peripheral blood samples. The mean and a 95% confidence interval will be calculated around the mean change from baseline.
Rate of recurrence (Phase I) | At approximately 3 months post treatment, and during long term followup will be part (every 3 to 6 months up to 3 years)
  Will be evaluated with standard-of-care CT and/or MRI to detect evidence of disease. The recurrence proportion and exact 95% confidence interval will be calculated.
Rate of local recurrence (Phase II) | Within 3 years post treatment during standard of care follow ups
  Will be assessed by standard-of-care CT and/or MRI. The recurrence proportion and exact 95% confidence interval will be calculated.
Disease free survival (Phase II) | Up to 3 years after treatment
  Will be detected via standard-of-care CT and/or MRI during the long-term follow-up that will be part of standard of care. The recurrence proportion and exact 95% confidence interval will be calculated.
Correlation between disease free survival and changes in levels of CEA (Phase II) | At 4-6 weeks after treatment
  Monitoring of CEA levels in correlation with disease free survival
Correlation between disease free survival and changes in levels of ctDNA (Phase II) | At 4-6 weeks after treatment
  Monitoring of ctDNA levels in correlation with disease free survival

CONTACTS AND LOCATIONS:
Overall Officials: Anthony S Dakwar, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States